CLINICAL TRIAL: NCT03993964
Title: A Multicenter, Phase II Open Label Study of Pyrotinib Maleate Combined With CDK4/6 Inhibitor SHR6390 in Treatment of HER2-positive Metastatic Breast Cancer
Brief Title: Study to Evaluate the Efficacy and Safety of CDK4/6 Inhibitor SHR6390 Combined With Pyrotinib in the Treatment of HER2-positive Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, wang shusen, clinical professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR-BLTN-014
Record Dates: First submitted 2019-06-13; First posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Pyrotinib + SHR6390 (Experimental): Pyrotinib combine with SHR6390 should be administrate to all subjects. pyrotinib 400mg qd combined with SHR 6390 125mg qd
  Interventions: Drug: Pyrotinib combine with SHR6390

INTERVENTIONS:
Drug: Pyrotinib combine with SHR6390 — SHR6390 is a novel small molecule inhibitor specifically targeting the CDK4/6 pathway. Pyrotinib is an irreversible pan-ErbB inhibitor which shows promising antitumour activity in patients with HER2-positive metastatic breast cancer

SUMMARY:
The main purpose of this study was to observe the efficacy and safety of treatment with pyrotinib and CDK4/6 inhibitor SHR6390 for HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Local recurrent or metastatic breast cancer suitable for chemotherapy, confirmed histologically.
* HER2-positive breast cancer(according to 2018 ASCO/CAP HER2 test guideline).
* Patients with HER2-positive metastatic breast cancer who had received ≤ 1-line treatment in the past;
* 18-70 years old.
* ECOG PS 0～1.
* life expectancy is not less than 12 weeks.
* at least one measurable lesion according to RECIST 1.1.
* ANC ≥ 2.0×109/L,PLT ≥ 100×109/L,Hb ≥ 90 g/L;TBIL≤1.5ULN；ALT and AST≤3×ULN（ALT and AST≤5×ULN if liver metastasis）;BUN and Cr≤1.5×ULN
* LVEF ≥ 50% and QTc≤470 ms.

Exclusion Criteria:

* Patients with symptomatic brain metastasis;
* Unable to swallow, chronic diarrhea and intestinal obstruction, there are many factors affecting drug use and absorption.
* patient who received radiotherapy, chemotherapy, surgery (excluding local puncture) or molecular targeted therapy within 4 weeks before admission; those who received anti-tumor endocrine therapy after screening period
* Participated in other drug clinical trials within 4 weeks before admission
* Tyrosine kinase inhibitors targeting HER2 (Neratinib, Lapatinib, pyrotinib, etc.) have been used or are being used in the past.
* Other malignant tumors, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma, have been diagnosed in the past five years.
* A history of immunodeficiency, including HIV positive, HCV,, or other acquired, congenital immunodeficiency disorders, or organ transplantation, is known.
* Has suffered from any heart disease
* Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial
* According to the judgement of the researchers, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of research (including, but not limited to, severe hypertension, severe diabetes, active infections, etc.).
* Moderate infection occurs within 4 weeks before the first administration (e.g. intravenous drip of antibiotics, antifungal or antiviral drugs according to clinical criteria), fever（> 38.5 ℃） of unknown origin occurs during the screening period/before the first administration.
* Researchers believe that patients are not suitable for any other situation in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-15 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | from enrollment to progression or death (for any reason), assessed up to 100 months
  CR+PR

SECONDARY OUTCOMES:
PFS | from enrollment to progression or death (for any reason),assessed up to 100 months
  Progression-Free Survival
OS | from enrollment to death (for any reason).assessed up to 100 months
  Overall Survival

IPD SHARING:
Plan to Share IPD: No